CLINICAL TRIAL: NCT04904523
Title: Project Sepsis: Blood Markers Including Molecular and Cellular Profiling for Identifying and Investigating Severe CoronaVirus Disease 2019 and Sepsis in Children and Young People (pSEP/COVID-ChYP)
Brief Title: Blood Markers for Identifying & Investigating Infection With COVID19 & Sepsis in Children.
Acronym: pSeP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiff University (Other)
Collaborators: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Other Study IDs: pSEP-COVID ChYP 263530
Record Dates: First submitted 2021-05-26; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Sepsis
MeSH Terms: conditions — COVID-19; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples will be collected, processed and RNA may be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases:
  1. Children and young people up to age 18 years, admitted to PCCU with probable or confirmed COVID-19, irrespective of severity of illness. This includes patients transferred from other hospitals as well as those admitted from Accident and Emergency department.
  Interventions: Diagnostic Test: Diagnostic Test:Blood test
- Controls: Controls:
  1. Children proven to have a non COVID infectious illness on laboratory testing.
  2. Children with sepsis or septic shock due to non-COVID infectious illness.
  3. Children or young people admitted to PCCU following accidental trauma.
  Interventions: Diagnostic Test: Diagnostic Test:Blood test

INTERVENTIONS:
Diagnostic Test: Diagnostic Test:Blood test — Drop of blood for RNA and metabolic analysis

SUMMARY:
Corona Virus Disease or COVID-19 is caused by SARS-CoV-2 virus. There have been reports of serious COVID-19 illness in children. In addition it has been linked to clusters of children presenting with high fevers and inflammation.

Sepsis, also called blood poisoning, is an abnormal response of the body to some infections. We aim to conduct research in children under 18 admitted to intensive care unit.

Using a systems approach towards mapping the body's immune and metabolic responses to COVID-19 or related illnesses and compare with other sepsis like illnesses.

DETAILED DESCRIPTION:
Corona Virus Disease or COVID-19 is caused by SARS-CoV-2 virus. There have been reports of serious COVID-19 illness in children. In addition it has been linked to clusters of children presenting with high fevers and inflammation.

Sepsis, also called blood poisoning, is an abnormal response of the body to some infections. We aim to conduct research in children under 18 admitted to intensive care unit and wards using blood samples. Blood samples as small as a quarter of a teaspoon, will be collected only alongside other routine blood tests. By analysing the blood samples, we aim to identify unique signals of information from the child or young person's genetic code as well as other chemical markers. This is to map the body's immune and metabolic response to COVID-19 or related illness and compare with other illnesses like sepsis. It will help us better understand COVID-19 illness and its association with the abnormal inflammatory response. The research will not delay emergency treatment for children or young people. Appropriate procedures for consent such as deferred consent will be used in children or young people with serious illness. Young people of 16 and 17 years of age will be assessed for capacity to consent. The study results will not influence the clinical care of patients. The research would not be identifying any other genetic disorders. Even though the data obtained includes some unique genetic information, the research only uses anonymised details from patients and there is no risk to confidentiality. Remaining blood following analysis will be stored in Biobank for an agreed duration. Specific consent will be obtained from parents or legal guardians, or young people with capacity for analysis and collection of unique genetic data, clinical information, sample storage and use of anonymous but unique genetic data for other research.

ELIGIBILITY:
Inclusion Criteria: Children or young people< 18 years who are admitted to PCCU and who have an acute illness are eligible for participation in the study.

Children and young people from age 0 day to <18 years with confirmed COVID-19 illness and/or those who meet the Multisystem inflammatory syndrome case definition.

-

Exclusion Criteria:

* Admitted to hospital for social reasons Or Declined consent by Parents or carers with legal responsibility or competent child Or Admitted to PCCU following a planned surgical procedure without an acute illness Or Direct clinical care team not able to provide research information in a language appropriate for non-English/Welsh speaking participants

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cases:
  1. Children and young people up to age 18 years, admitted to PCCU with probable or confirmed COVID-19, irrespective of severity of illness. This includes patients transferred from other hospitals as well as those admitted from Accident and Emergency department.
  Controls:
  1. Children proven to have a non COVID infectious illness on laboratory testing.
  2. Children with sepsis or septic shock due to non-COVID infectious illness.
  3. Children or young people admitted to PCCU following accidental trauma.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Outcome 1 | 3 years
  To evaluate known blood molecular and genomic markers of infection in children and young persons with confirmed or probable COVID19 and compare with non COVID19 illnesses.

SECONDARY OUTCOMES:
Outcome 2 | 3 Years
  To investigate systemic pathway biology of SARS-CoV-2 infection and by comparison with other viral and bacterial sepsis cases identify new signatures associated with COVID-19 in patients up to 18 years of age.
  To profile molecular analytes (proteins, lipids and nucleic acids) and blood cell phenotypes in children with sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiff University, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oruganti S, Rodrigues PRS, White D, Watkins WJ, Shapey S, Barrow A, Al Samsam R, Ali S, Gajraj M, Skone R, Jardine M, Evans J, Struik S, Song JE, Abood L, Paquete B, Foulkes S, Saunders B, Strang A, Kotecha SJ, Phillips B, Evans A, Buchanan I, Bowes S, Ali B, Gore M, Thomas-Turner R, Andrews R, Zaher S, Sharma S, Chakraborty M, Parkinson E, Liberatore F, Woolley T, Edkins S, Davies LC, Moet L, McLaren JE, Watson GL, O'Donnell V, Hood K, Ghazal P. Immune and metabolic markers for identifying and investigating severe Coronavirus disease and Sepsis in children and young people (pSeP/COVID ChYP study): protocol for a prospective cohort study. BMJ Open. 2023 Mar 27;13(3):e067002. doi: 10.1136/bmjopen-2022-067002. PMID 36972964